CLINICAL TRIAL: NCT03924271
Title: Prevalence Study of Iron Deficiency in Patients With Cancer
Acronym: CARENFER ONCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARENFER ONCO HEMATO
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONCOLOGY (Experimental): Patient with a cancer
  Interventions: Diagnostic Test: Iron deficiency testing

INTERVENTIONS:
Diagnostic Test: Iron deficiency testing — Blood sample for complete iron status

SUMMARY:
Despite its high prevalence, a recent study conducted by Prof. Cacoub (unpublished) on the french national health insurance database showed that iron deficiency was an underdiagnosed and under-treated co-morbidity. In inflammatory situations, especially during cancer, the measurement of the transferrin saturation factor is only performed in about 10% of cases whereas this measure is recommended in inflammatory situations including cancer (French Health High Authority 2011)

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over the age of 18
* Patient in an oncology department (any type of tumor, any type of treatment, initiated or not)
* Patient affiliated or beneficiary of a social security system
* Patient with written consent

Exclusion Criteria:

* Protected patient: major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2019-05-15 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood iron status | One day
  ferritin, haemoglobin, transferrin saturation factor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luporsi E, Turpin A, Massard V, Morin S, Chauffert B, Carnot A, Cacoub P; Behalf of the CARENFER Study Group. Iron deficiency in patients with cancer: a prospective cross-sectional study. BMJ Support Palliat Care. 2024 May 17;14(2):215-221. doi: 10.1136/bmjspcare-2021-002913. PMID 34330792